CLINICAL TRIAL: NCT00128479
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Safety and Efficacy of Three Dose Levels of CORLUX™ (Mifepristone) Plus an Antidepressant vs. Placebo Plus an Antidepressant in the Treatment of Psychotic Symptoms in Patients With Major Depressive Disorder With Psychotic Features (PMD)
Brief Title: A United States Study of the Safety and Tolerability of Corlux for Psychotic Symptoms in Psychotic Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-1073-06
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Major Depressive Disorder; Psychotic Disorders
Keywords: PMD; Psychotic Depression; Psychosis; Major Depression; Depression; Psychotic Major Depression
MeSH Terms: conditions — Depressive Disorder, Major; Psychotic Disorders; Depression | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- mifepristone 300 mg (Experimental)
  Interventions: Drug: mifepristone
- placebo (Placebo Comparator)
  Interventions: Drug: mifepristone matched placebo
- mifepristone 600 mg (Experimental)
  Interventions: Drug: mifepristone 600 mg
- mifepristone 1200 mg (Experimental)
  Interventions: Drug: mifepristone 1200 mg

INTERVENTIONS:
Drug: mifepristone — mifepristone 300 mg daily for 7 dats
  Arms: mifepristone 300 mg
Drug: mifepristone matched placebo — daily for 7 days
  Arms: placebo
Drug: mifepristone 600 mg — mifepristone 600 mg daily for 7 days
  Arms: mifepristone 600 mg
Drug: mifepristone 1200 mg — mifepristone 1200 mg daily for 7 days
  Arms: mifepristone 1200 mg

SUMMARY:
Corlux (mifepristone) is a new medication that modulates the body's use of a hormone called cortisol. Under normal conditions, cortisol and other hormones are created by the body in response to physical and emotional stress, triggering a healthy stress response. People who suffer from psychotic major depression may have unusually high levels of cortisol circulating within them or abnormal patterns of cortisol levels, overloading the stress response mechanism and causing symptoms of psychosis such as delusional thoughts or hallucinations. If Corlux can keep the body's cortisol receptors from being overloaded, the stress response system may return to normal function, which may result in improvement of symptoms. The purpose of this 56 day study is to learn the safety and effectiveness of Corlux in patients who have been diagnosed with psychotic major depression (PMD).

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for enrollment into this study are male and female adult patients who:

* Are 18 to 75 years of age
* Have a diagnosis of major depressive disorder with psychotic features (DSM-IV 296.24 or 296.34)
* Are able to provide written informed consent.

Exclusion Criteria:

Individuals not eligible to be enrolled into the study are those who:

* Have a major medical problem
* Have previously participated in a CORLUX (C-1073, mifepristone) clinical trial
* Have a history of an allergic reaction to CORLUX (C-1073, mifepristone).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2004-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The change in a measure of psychosis | screen, Days 0, 7, 14, 28, 42, 56

SECONDARY OUTCOMES:
The change in a measure of depression | screen, Days 0,7, 14, 28, 42, 56

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Beebe, PhD, Study Director — Corcept Therapeutics
Locations (44):
- United States (44):
  - K&S Research Services, Little Rock, Arkansas
  - Center for Emotional Fitness, Cerritos, California
  - Harbor Medical Associates, Inc., Fountain Valley, California
  - Synergy Clinical Research Center, National City, California
  - Excell Research, Oceanside, California
  - Pacific Clinical Research Medical Group, Riverside, California
  - AV Institute, Inc., Torrance, California
  - Neuropsychiatric Institute of Orange County, Westminster, California
  - Geriatric and Adult Psych, Hamden, Connecticut
  - Comprehensive NeuroScience, Inc., Washington D.C., District of Columbia
  - Professional Clinical Research Inc., Fort Lauderdale, Florida
  - Amit Vijapura, MD, Jacksonville, Florida
  - Tukoi Inst for Clinical Research, Miami, Florida
  - Bioquan Research Group, Inc., North Miami, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Mark Ashby, MD, Sebring, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Hawaii Clinical Research Center, Honolulu, Hawaii
  - Midwest Center for Neurobehavioral Medicine, Oakbrook Terrace, Illinois
  - Peryam and Kroll Health Care Research, Schaumburg, Illinois
  - Clintell, Inc., Skokie, Illinois
  - CTT Research, Prairie Village, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Louisiana Research Associates, Inc, New Orleans, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Saaid Khojasteh & Assoc, Inc, Saint Charles, Missouri
  - Medex Healthcare Research, St Louis, Missouri
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Brooklyn Medical Institute, Brooklyn, New York
  - Advanced Bio-Behavioral Science, Inc, Elmsford, New York
  - Saint Vincent Catholic Medical Centers of New York, Staten Island, New York
  - Anxiety and Depression Clinic at Montefiore Medical Center, The Bronx, New York
  - Lutheran Hospital, Cleveland, Ohio
  - Southwest Cleveland Sleep Center, Inc., Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Crossroads Counseling & Consulting Associates, Moon Township, Pennsylvania
  - CNS Research Institute (CRI), Philadelphia, Pennsylvania
  - Segal Institute, Charleston, South Carolina
  - Harmony Research, Johnson City, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - The Cedars Hospital, InSite Clinical Research, DeSoto, Texas
  - Felin-Jennings Clinic, Houston, Texas
  - R&D Clinical Research, Inc., Lake Jackson, Texas
  - America's Doctor/Essential Doctor, Inc, Seattle, Washington

REFERENCES:
- [Background] Brogden RN, Goa KL, Faulds D. Mifepristone. A review of its pharmacodynamic and pharmacokinetic properties, and therapeutic potential. Drugs. 1993 Mar;45(3):384-409. doi: 10.2165/00003495-199345030-00007. PMID 7682909
- [Background] Belanoff JK, Rothschild AJ, Cassidy F, DeBattista C, Baulieu EE, Schold C, Schatzberg AF. An open label trial of C-1073 (mifepristone) for psychotic major depression. Biol Psychiatry. 2002 Sep 1;52(5):386-92. doi: 10.1016/s0006-3223(02)01432-4. PMID 12242054
- [Background] Belanoff JK, Flores BH, Kalezhan M, Sund B, Schatzberg AF. Rapid reversal of psychotic depression using mifepristone. J Clin Psychopharmacol. 2001 Oct;21(5):516-21. doi: 10.1097/00004714-200110000-00009. PMID 11593077
- [Derived] Kruizinga J, Liemburg E, Burger H, Cipriani A, Geddes J, Robertson L, Vogelaar B, Nolen WA. Pharmacological treatment for psychotic depression. Cochrane Database Syst Rev. 2021 Dec 7;12(12):CD004044. doi: 10.1002/14651858.CD004044.pub5. PMID 34875106
- [Derived] Block TS, Kushner H, Kalin N, Nelson C, Belanoff J, Schatzberg A. Combined Analysis of Mifepristone for Psychotic Depression: Plasma Levels Associated With Clinical Response. Biol Psychiatry. 2018 Jul 1;84(1):46-54. doi: 10.1016/j.biopsych.2018.01.008. Epub 2018 Jan 31. PMID 29523415
- See also: Corcept Therapeutics — http://www.corcept.com